CLINICAL TRIAL: NCT04206826
Title: Tolerance and Efficiency of an Intrabuccal Biological Film to Enhance Oral Dryness Sensation: The "PREDELFI" Clinical Pilot Study
Acronym: PREDELFI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 29BRC18.0037 (PREDELFI)
Record Dates: First submitted 2019-12-10; First posted 2019-12-20 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2021-05

CONDITIONS: Sicca Syndrome; Xerostomia
Keywords: natural film; prebiotics
MeSH Terms: conditions — Sjogren's Syndrome; Xerostomia

STUDY DESIGN:
Intervention Model Description: Each patient will apply the two films (PreDelfi and control according to randomization) at the level of the gingival mucosa next to the maxillary vestibule for 30 days
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PREDELFI Film (Experimental)
  Interventions: Device: PREDELFI
- CONTROL Film (Placebo Comparator)
  Interventions: Device: CONTROL

INTERVENTIONS:
Device: PREDELFI — It's a natural film which contains a concentrated alpha-GOS (alpha-galacto-oligosaccharide) soy extract, a milk protein concentrate containing caseins and whey proteins and vegetable glycerin
  Arms: PREDELFI Film
Device: CONTROL — It's a natural film which is devoided of active ingredient. It contains sodium alginate; vegetable glycerin, caramel, beta carotene and water.
  Arms: CONTROL Film

SUMMARY:
Xerostomia affects at least a quarter of the population. This prevalence is increased in postmenopausal women and people over 65 years of age. Associated with age are systemic diseases such as Sjögren's Syndrome, diabetes, Parkinson's disease or cancer. It handicaps the patient in his social life, but also in terms of his well-being by the consequences it generates in the oral cavity. This dryness may be the consequence of taking certain medications, head and neck radiotherapy, but also being a symptom of an underlying pathology whose screening will allow early treatment and avoid complications. Today, no single therapeutic solution is enough and patients are waiting for new therapeutic innovations in this area. This study proposes to evaluate the tolerance of an adhesive film containing prebiotics by comparing it to a placebo control film.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the tolerance of an adhesive film containing prebiotics on the improvement of signs and symptoms related to dry mouth by comparing it to a placebo film.

The primary endpoint is the assessment of tolerability assessed using a visual analogue scale (VAS) from 0 to 100 at the end of the 1-month period of both treatment periods (D30 and D90). In this study, the efficacy and tolerance of the adhesive film containing prebiotics will be analyzed.

Each participant in this study will receive two galenic forms of the medical device whose allocation order was previously defined by a randomization list.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 18 or over
* Complaining of xerostomia and validated by a standardized question
* With hyposialia diagnosed by the measurement of stimulated salivary flow (DSS) and unstimulated (DNS)
* Patient having signed a consent
* Registered with Social Security

Exclusion Criteria:

* The patient having known sensitivity to any of the products or components of the biofilms (milk protein, soy derivatives, sodium alginate, vegetable glycerin, caramel and beta carotene)
* Allergic to birch and / or peanut
* Having an ethyl intoxication (> 2 glasses of wine / day), smoking (> 10 cigarettes / day)
* Unable to complete self-assessment questionnaires or to follow study protocol procedures (unable to read and / or write).
* Participant in another clinical study at the time of inclusion or having participated in the 30 days preceding recruitment in this study
* Having a life-threatening condition for the duration of the study
* Treated with sialogogues (pilocarpine hydrochloride) within 30 days prior to inclusion
* Using salivary substitutes
* Protected persons within the law (articles L1121-5 to L1121-8)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-06-25 (Actual); Primary Completion 2021-04-23 (Actual); Study Completion 2021-04-23 (Actual)

PRIMARY OUTCOMES:
Tolerance evaluation | day 90
  The primary endpoint is a composite endpoint of tolerance evaluation defined by:
  * the patient (EVA from 0 to 100),
  * the investigator (degree of redness and inflammation of the mucous membranes opposite the site of the device,
  * reporting adverse events related to the device

SECONDARY OUTCOMES:
Oral comfort | day 90
  Self-evaluation of the patient's oral dryness (oral comfort) using a 100mm visual analogue scale (measurement of the absolute variation at the beginning and end of each treatment period)
Subjective evaluation of dry mouth | day 90
  Subjective evaluation of the absolute variation of the specific signs and symptoms of dry mouth (difficulty speaking, chewing swallowing, taste alteration, burning sensations) using 100 mm analogue visual scales
Clinical assessment of the mucous | day 90
  Objective clinical assessment of the general condition of the mucous membranes (redness, dryness, degree of inflammation of periodontal tissues, mucous membranes,...)
Evaluation of salivary flow | day 90
  Objective evaluation of the absolute variation of the stimulated and unstimulated salivary flow rates according to the dosage forms used and the variation of the oral pH using specific strips.
Evaluation of the salivary microbiota | day 90
  Evaluation by molecular sequencing of the salivary microbiota to study the impact of the film on the modification of the salivary microbiota (quantification of the different species by NGS)

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning five years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.

REFERENCES:
- [Derived] Orliaguet M, Fong SB, Le Pottier L, Meuric V, Boisrame S, Bonnaure-Mallet M, Pers JO. Tolerance to intraoral biofilms and their effectiveness in improving mouth dryness and modifying oral microbiota in patients with primary Sjogren's syndrome: "Predelfi study". Front Microbiol. 2023 Feb 8;14:1071683. doi: 10.3389/fmicb.2023.1071683. eCollection 2023. PMID 37293235